CLINICAL TRIAL: NCT03411720
Title: Whole Body Exercise in Spinal Cord Injury: Effects on Psychosocial Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Collaborators: The Craig H. Neilsen Foundation (Other)
Responsible Party: Principal Investigator, J. Andrew Taylor, Director, Cardiovascular Research Laboratory, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2017D006049
Record Dates: First submitted 2018-01-05; First posted 2018-01-26 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FES-row-training (Experimental): Subjects will perform 4 months of FES-row-raining
  Interventions: Other: FES Row Training
- Wait-list time control (Other): Subjects will wait 4 months before performing being allowed to engage in 4 months of FES-row-training
  Interventions: Other: FES Row Training
- Arms-only-row-training (Active Comparator): Subjects will perform 4 months of arms-only row training before being allowed to engage in 4 months of FES-row-training
  Interventions: Other: FES Row Training

INTERVENTIONS:
Other: FES Row Training — Hybrid FES Row Training using voluntary upper body and electrically-stimulated lower body

SUMMARY:
Persons with spinal cord injury (SCI) are confronted with a multitude of psychological and physiological changes post-injury leading to seemingly insurmountable barriers to participating in daily life. After injury persons with SCI engage in fewer social interactions, spend more time sedentary, and are less likely to leave the home. This leads to restricted social participation that, in turn, contributes to greater psychological problems and negatively impacts the lives of adults with SCI. Intense, structured exercise has substantial potential benefits for improving psychosocial wellbeing among persons with SCI, but accessible exercise options are few and cannot achieve high intensities of whole-body exercise. This work will use approaches to overcome the barriers to intense exercise. The investigators will use hybrid functional electrical stimulation row training (FESRT) to allow for a more intense exercise stimulus, potentially having a greater impact on psychosocial wellbeing. There is initial evidence that persons with mobility impairments who are highly physically active demonstrate better psychosocial wellbeing compared with those who have low levels of physical activity. A limitation to understanding the influence of exercise on psychosocial wellbeing is the lack of robust and time-dependent measures. The investigators will use a smartphone-based research application to measure psychosocial well-being, thus decreasing self-report bias and capturing in-the-moment behavioral and self-report data.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18 years of age)

  * Be in good health (asymptomatic for acute treatable illness) and medically cleared to exercise
  * Own an iPhone or Android smartphone with the capacity to download and run the research platform (able to log into to the relevant app store, install the app on their own phone, and run the app).
  * Be able to understand, communicate with and be understood by research personnel or Interpreters
  * Be interested in participating and provide informed consent
  * Have a SCI with motor or sensory deficits and use a wheelchair as primary means of mobility
  * Have an injury level only as high as C4 to allow sufficient arm function for rowing

Exclusion Criteria:

* Participants will not have previously completed FESRT
* Acute illness
* Musculoskeletal injuries that have not healed completely
* Had heart surgery or are status post-myocardial infarction (MI) in the last 4 to 6 months, -Unstable angina
* Uncontrolled hypertension (systolic blood pressure ≥160 mm Hg and/or diastolic blood pressure ≥100 mm Hg)
* uncontrolled dysrhythmias
* Recent history of congestive heart failure that has not been evaluated and effectively treated
* Severe stenotic or regurgitant valvular disease
* Hypertrophic cardiomyopathy
* Unhealed pressure ulcer Stage 2 or higher at relevant contact sites during exercise.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Depression | Each week during the 4 months
  Difference between groups in depression symptom severity (Patient Health Questionnaire-9); Within-individual Correlation of exercise intensity with depression
Pain Severity | Each week during the 4 months
  Difference between groups in pain severity, rated on a 0-10 scale ("0 being no pain and 10 being pain so severe you couldn't stand it"); Within-individual Correlation of exercise intensity with pain.
Pain Interference | Each week during the 4 months
  Difference between groups in pain interference in daily life activities ("0. Not at all 1. A little bit 2. Moderately 3. Quite a bit 4. Extremely"); Within-individual Correlation of exercise intensity with pain.
Anxiety | Each week during the 4 months
  Difference between groups in anxiety (Spinal Cord Injury Quality of Life Anxiety Short Form); Within-individual Correlation of exercise intensity with anxiety. Minimum score is 9, Maximum score is 45. Higher scores indicate higher anxiety.
Satisfaction with Social Participation | Each week during the 4 months
  Difference between groups in satisfaction with social roles and activities (Spinal Cord Injury Quality of Life Satisfaction with Social Roles and Activities Short Form); Within-individual Correlation of exercise intensity with satisfaction with social participation. The Minimum score is 20 and the maximum score is 50. Higher values indicate greater satisfaction with social participation.
Ability to participate in social roles | Each week during the 4 months
  Difference between groups in ability to participate in social roles and activities. Spinal Cord Injury Quality of Life Ability to Participate in Social Roles and Activities Short Form. Within-individual Correlation of exercise intensity with ability to participate in social roles. The Minimum score is 20 and the maximum score is 50. Higher values indicate greater satisfaction with social participation.

SECONDARY OUTCOMES:
Health Complications | Each week during the 4 months
  Difference between groups in frequency of secondary health complications; Within-individual Correlation of exercise intensity with secondary health complications.
Community Mobility | Each week during the 4 months
  Difference between groups in community mobility (Distance traveled each week); Within-individual Correlation of exercise intensity with community mobility.
Social Connectivity: Frequency | Each week during the 4 months
  Difference between groups in social connectivity (Frequency of phone calls and text messages); Within-individual Correlation of exercise intensity with frequency of social connectivity.
Social Connectivity: Reciprocity | Each week during the 4 months
  Difference between groups in social connectivity (Reciprocity of phone calls and text messages); Within-individual Correlation of exercise intensity with reciprocity of social connectivity.

CONTACTS AND LOCATIONS:
Overall Officials: J. Andrew Taylor, Principal Investigator — Spaulding Rehabilitation Hospital/Harvard Medical School
Locations (1):
- Spaulding Rehabilitation Network, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No